CLINICAL TRIAL: NCT02144116
Title: Effects of a Dance-movement Therapy Programme in Patients With Fibromyalgia.
Brief Title: Dance-movement Therapy Programme in Fibromyalgia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Proffesor assistant, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0052UG
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Fibromyalgia
Keywords: dance-movement therapy; balance; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Methods; Dance Therapy; Occupational Therapy; Control Groups; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Patients with fibromyalgia included in a dance-movement therapy programme
  Interventions: Other: Dance-movement therapy
- Control group (Active Comparator): Patients with fibromyalgia who receive a standardized educational information in the form of a leaflet about balance disorders and quality of life in fibromyalgia.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Dance-movement therapy — The dance-movement was practised in groups. Dance-movement therapy derived from dance education. The goals of dance-movement therapy included assessing patient needs, communicating emotions, improving self-control, organizing thoughts and actions, developing interpersonal skills, integrating physical and emotional selves, promoting body awareness, and supporting healing.
  Other Names: intervention; dance therapy; occupational therapy
  Arms: Experimental group
Other: Control group — Standardized educational information in the form of a leaflet about balance disorders and quality of life in fibromyalgia.
  Other Names: Control; Education
  Arms: Control group

SUMMARY:
Fibromyalgia is a chronic illness characterized by persistent widespread muscle pain with generalized hyperalgesia and allodynia. It can be accompanied by other concomitant symptoms like fatigue, sleep disturbances, musculoskeletal disorders, distress and psychological disorders. This condition is very prevalent. It has been reported to be about 2-5% of the general global population. Fibromyalgia is associated with balance problems and increased fall frequency. The objective of this study was to examine the effects of an 8 weeks dance-movement therapy programme on balance, strength, flexibility and quality of life in patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic condition associated with balance problems and pain. It has been previously described that fibromyalgia may affect peripheral and/or central mechanisms of postural control. Balance or postural stability is a very complex task that involves the integration of multiple sensory inputs to execute appropriate neuromuscular activity needed to maintain balance.

Patients with fibromyalgia have also muscle weakness. Muscle strength depends on both the cross-sectional area of the muscle and the neural activity. Range of movement and quality of life have also been reported to be affected.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed of Fibromyalgia attending to the Fibromyalgia Association of Granada.
* Women who can complete the assessment battery of tests at the beginning and at the end of the study

Exclusion Criteria:

* Auditive and visual disturbances.
* Cognitive problems.
* Psychiatric pathology.
* Traumatic pathology of lower limbs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Changes in balance | Baseline, 8 weeks
  Balance is going to be assessed with the Mini BalanceEvaluation System Test. This test assesses dynamic balance, with four subscales:anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait.
  The Mini BESTest is a 14 item test scored on a 3 level ordinal scale. For the Mini BESTest, the original BESTest 4 level (0 - 3) scoring was revised to 3 levels (0 - 2) due to redundancy. Total score = 28 points per test directions. Two items have right and left assessment in which the lower score is used within the total score (directions specify which to use). For research, many studies specify use of both left and right data, thus calculating data based on 32 (vs 28) points

SECONDARY OUTCOMES:
Changes in quadriceps strength | Baseline, 8 weeks
  Changes from baseline to postintervention on quadriceps strength. This will be measured using a Jamar dynamometer with a standard protocol allowing three attempts on each side. The maximum value achieved from all six attempts was used in analyses. Kg/cm2.
Changes in quality of life | Baseline, 8 weeks
  Quality of life associated with health. This is going to be measure with the EuroQol-5 questionnaire.
Changes in flexibility of lower limbs | Baseline, 8 weeks
  Changes from baseline to postintervention measured with neurodynamic tests It is going to be measured with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided